CLINICAL TRIAL: NCT00758797
Title: In Situ Photoimmunotherapy: A Tumor Directed Treatment for Advanced Melanoma With Cutaneous Metastases
Brief Title: A Novel Treatment for Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was not renewed during annual Northwestern Cancer Center review.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU1213
Record Dates: First submitted 2008-06-23; First posted 2008-09-25 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Melanoma
Keywords: metastatic melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): DIOMED laser + photosensitizing agent injected intralesionally and topical immuno-modulating cream
  Interventions: Other: Photoimmunotherapy

INTERVENTIONS:
Other: Photoimmunotherapy — DIOMED laser + photosensitizing agent injected intralesionally and topical immuno-modulating cream

SUMMARY:
A novel treatment for metastatic melanoma combining a laser and an immune-system stimulating cream.

DETAILED DESCRIPTION:
A novel treatment for metastatic melanoma combining a laser and an immune-system stimulating cream with or without injection of a substance that makes the tumor more sensitive to the laser.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Subjects must have Stage III or IV melanoma with histologically confirmed cutaneous metastatic malignant melanoma from any tumor site.
3. Subjects must have measurable disease. See section 10.2 for the evaluation of measurable disease (RECIST).
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
5. Required laboratory parameters (all blood tests must be obtained within 14 days prior to the start of the study treatment):

Platelet count > 40,000 per mm3 Absolute Neutrophil Count (ANC) > 1,500 per mm3

Exclusion Criteria:

1. Life expectancy, in the opinion of the investigator of less than 4 months
2. Known allergy to any drugs used in treatment
3. Immunosuppression, including HIV positive subjects, use of systemic steroids daily or other immunosuppressive medications within 1 month of treatment
4. Chemotherapy/immunotherapy within 4 weeks of initiation
5. Local chemotherapy or immunotherapy to target lesions with 4 weeks of initiation
6. Radiation therapy at the treatment site within 4 weeks of initiation
7. Uncontrolled brain metastases
8. History of cutaneous photosensitization or photodermatoses
9. Non-treated, active cancers other than melanoma and non-melanoma skin cancers.
10. Active infectious disease requiring antibiotic therapy
11. Unstable medical illness
12. Past or present major psychiatric illness
13. Pregnant or lactating women
14. End stage renal disease or serum creatinine greater than the upper limit of normal or creatinine clearance <50cc/min
15. Acute hepatitis (any cause)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Tolerability, safety, toxicity, of novel treatment through evaluation of subject response and physician observation of adverse events. | 24 weeks

SECONDARY OUTCOMES:
Assess time to disease progression | 24 weeks to years
Evaluate tumor response by measuring clinically apparent tumors throughout study. | 24 weeks
Quantify overall survival in this study population | years

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States